CLINICAL TRIAL: NCT00442494
Title: Feasibility of Corticosteroid in the Prevention of Atrial Fibrillation After Cardiac Surgery: A Prospective, Double-Blind Randomized Multicenter Trial
Brief Title: Corticosteroids for the Prevention of Atrial Fibrillation After Cardiac Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has been completed as planned
Sponsor: Kuopio University Hospital (Other)
Collaborators: Tampere University Hospital (Other); Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Helena Pehkonen, assistant, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: KUH5204515
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-10

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation after cardiac surgery
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study couldn´t start due to investigator (Other): Study couldn´t start due to investigator
  Interventions: Drug: intravenous hydrocortisone

INTERVENTIONS:
Drug: intravenous hydrocortisone

SUMMARY:
Atrial fibrillation is the most common arrhythmia to occur after cardiac surgery. Inflammatory response may be one etiological factor.

We hypothesized that intravenous corticosteroid administration after cardiac surgery prevents AF after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo their first on-pump CABG, aortic valve replacement or combined aortic valve replacement and CABG were enrolled.

Exclusion Criteria:

* Previous episodes of AF or flutter
* Uncontrolled diabetes mellitus
* Systemic mycotic infection
* Active tuberculosis
* Cushing's syndrome
* Psychotic mental disorder
* Herpes Simplex keratitis
* Serum creatinine exceeding 200 µg/ml
* Patients were also excluded if they had a history of previous peptic ulcer or thrombophlebitis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Study couldn´t start due to investigator | Study couldn´t start due to investigator
  Study couldn´t start due to investigator

SECONDARY OUTCOMES:
Study couldn´t start due to investigator | Study couldn´t start due to investigator
  Study couldn´t start due to investigator

OTHER OUTCOMES:
Study couldn´t start due to investigator | Study couldn´t start due to investigator
  Study couldn´t start due to investigator

CONTACTS AND LOCATIONS:
Overall Officials: Jari Halonen, MD, Principal Investigator — Kuopio University Hospital

REFERENCES:
- [Derived] Voltarelli JC, Couri CE, Stracieri AB, Oliveira MC, Moraes DA, Pieroni F, Coutinho M, Malmegrim KC, Foss-Freitas MC, Simoes BP, Foss MC, Squiers E, Burt RK. Autologous nonmyeloablative hematopoietic stem cell transplantation in newly diagnosed type 1 diabetes mellitus. JAMA. 2007 Apr 11;297(14):1568-76. doi: 10.1001/jama.297.14.1568. PMID 17426276
- [Derived] Halonen J, Halonen P, Jarvinen O, Taskinen P, Auvinen T, Tarkka M, Hippelainen M, Juvonen T, Hartikainen J, Hakala T. Corticosteroids for the prevention of atrial fibrillation after cardiac surgery: a randomized controlled trial. JAMA. 2007 Apr 11;297(14):1562-7. doi: 10.1001/jama.297.14.1562. PMID 17426275